CLINICAL TRIAL: NCT03613389
Title: Prevention of Oral Mucositis After Using Oral Topical Vitamin E Versus Voriconazole and Levofloxacin in Pediatric Cancer Patients Receiving Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Samah omer Mekki, B.D.S, Faculty of Dentistry, Khartoum College of Medical Sciences, Sudan (2011), Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CEBD-CU-2018-06-20
Record Dates: First submitted 2018-07-18; First posted 2018-08-03 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Oral Mucositis (Ulcerative) Due to Antineoplastic Therapy
MeSH Terms: conditions — Stomatitis; Ulcer | interventions — Vitamin E

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral topical vitamin E (Experimental)
  Interventions: Dietary Supplement: oral topical vitamin E
- voriconazole and levofloxacin (No Intervention)

INTERVENTIONS:
Dietary Supplement: oral topical vitamin E — Vitamin E is an antioxidant agent which may limit tissue damage from free oxygen radicals and, thus, may reduce the severity of mucositis during cancer treatments and protect cell membranes from radiation damage (Alterio et al., 2007). It has a very low toxicity and is generally well-tolerated (Geeraert et al., 2015).
  Arms: oral topical vitamin E

SUMMARY:
Statement of problem Oral mucositis is an inflammatory condition that affects mucosa of the oral cavity. The etiology of this kind of aggravation is related to the introduction of radiotherapy or chemotherapeutic medications. (Alvarino et al., 2014, Rohani et al., 2015) With the prevalence of mucositis up to 80% in pediatric patient (Cheng et al., 2004).

Clinically, oral mucositis is a painful situation that significantly affects patients' quality of life. The severe cases are associated with ulcerated mucosa and secondary infection which may led to life-threatening sepsis. (Kolokythas , et al., 2010) Oral mucositis is one of the most debilitating complications following chemotherapy, its remains an unresolved clinical problem, and it has physical and psychosocial implications for patients. The ulcerative lesions are often very painful, requiring treatment with analgesics and supportive nutrition, and the cancer treatment may need to be interrupted or modified. All these conditions may increase treatment costs, preclude further treatment and alter the quality of life of the patient. (Sonis et al., 2001) There are many oral care regimens including prophylactic antibacterial and antifungal drugs, Levofloxacin is antibacterial drug causing inhibition of cell wall synthesis agent, Levofloxacin failed to show any significant difference in mucositis or oral ulceration (Bucaneve et al., 2005). While voriconazole is antifungal that has been noted to cause transient visual disturbances and A major drawback is potential interactions with certain chemotherapy agents (Marks et al., 2011).

Vitamin E is an antioxidant agent which may limit tissue damage from free oxygen radicals and, thus, may reduce the severity of mucositis during cancer treatments and protect cell membranes from radiation damage (Alterio et al., 2007). It has a very low toxicity and is generally well-tolerated (Geeraert et al., 2015).

Rationale

There is no enough studies about vitamin E effect in reduction of oral mucositis.

El -Housseiny et al., (2007), recommend that oral mucositis is successfully treated by the topical application of vitamin "E", compared to its systemic administration. Vitamin "E" alone is not enough for the treatment of infected lesions; further studies using vitamin "E" to treat the infected lesions are needed.

Also based on the recommendation of Wadleigh et al., (1992) who was the first one to study the topical effect of vitamin "E" on oral mucositis; however, they did not know whether the effect was due to the topical application or the systemic absorption of the vitamin when applied topically.

Benefit to patient and population:

The vitamin E is nontoxic, odorless, tasteless, and well tolerated by the patients, reduce nutritional compromise, maintain impact on quality of life, and reasonable economic costs.

Benefits of practitioners and clinicians:

The use of vitamin E is easy to apply, not technique sensitive and it is cheap and readily available reducing clinical time.

DETAILED DESCRIPTION:
Title Prevention of oral mucositis after using oral topical vitamin E versus voriconazole and levofloxacin in pediatric cancer patients receiving chemotherapy.

Title registration:

The study is to be registered on ClinicalTrials.gov/

Protocol version:

Version (1)

Funding:

Self-funding Roles and responsibilities

Principle investigator:

Samah omer Mekki B.D.S, Faculty of Dentistry, Khartoum College of Medical Sciences, Sudan (2011) Will make case selection, methodology, instructions and patient recall. Then write the thesis and perform a master table for the results.

Main supervisor: Prof.Dr. Mahmoud Hamdy.

* Professor of Pediatric Dentistry and Dental Public Health, Faculty of Dentistry, Cairo University.
* Prof.Dr. Mahmoud Hamdy will supervise all procedures and sort out any foreseen or existing problem. He will initially consult with a statistician for developing the study design, statistical analysis, results presentation design and interpretation.

Assistant supervisor: Dr. Nada Wassef.

* Lecturer of Pediatric Dentistry and Dental Public Health, Faculty of Dentistry, Cairo University.
* The assistant supervisor will supervise clinical steps and findings revise and edit the draft of thesis.

Assistant supervisor: Dr. Asmaa Mohammed Hamoda

* Lecturer of Pediatric oncology, National cancer institute, Cairo university.
* Will validate diagnosis of selected cases to ensure that only indicated case are included in the study, clinical evaluation of post intervention findings and follow up. Revise, edit the first draft of thesis.

Trial sponsor:

Department of Pediatric oncology, National Cancer Institute, Cairo university.

Role of study sponsor:

Provide access to children receiving Chemotherapy.

Committees:

National Cancer Institute Committees:

1- Research Plan committee. 2- Department Board committee. 3-Ethics Committee. 4-Institute Board.

Department of Pediatric Dentistry, Faculty of Dentistry- Cairo University:

1. Department Board.
2. Research Plane Committee.
3. Evidence Based Committee, Faculty of Dentistry - Cairo University.
4. Ethics Committee, Faculty of Dentistry - Cairo University.
5. Higher Education and Research Committee.
6. Faculty Board.

   Research question:

   Is topical oral vitamin E application more effective in prevention of oral mucositis in pediatric cancer patients receiving chemotherapy compared to Voriconazole and Levofloxacin as standard protocol? Choice of comparators Aim of The Study The aim of the present study is to assess the prevention of oral mucositis after using oral topical vitamin E versus voriconazole and levofloxacin in pediatric cancer patients receiving chemotherapy.

   Hypothesis Objectives of The Study

   • Primary objective: To evaluate the Effectiveness of Vitamin E versus Voriconazole and Levofloxacin in prevention of chemotherapy induced oral mucositis in pediatric cancer patients.

   • Secondary objective: To evaluate the role of Vitamin E in prevention of chemotherapy induced oral mucositis in pediatric patients with cancer.

   Trial design:

   - A Randomized clinical trial.

   PICOS (P) Population: Children with cancer receiving chemotherapy. (I) Intervention: Topical vitamin "E" application. (C) Control: Voriconazole and Levofloxacin application. (O) Outcome: Outcome measure Outcome measuring Outcome measuring unit

   Primary outcome:

   Patient reported mucositis Children's International Mucositis Evaluation Scale (ChIMES). (Jacobs et al., 2013) (Appendix A)

   Score (0-5)

   Secondary outcome:

   Clinical assessment of mucositis Oral mucositis WHO Toxicity System (Dos Reis et al., 2016) (Appendix B) Score (0-4)

   - Study (S): A Randomized clinical trial.

   Search strategy:

   - Keywords: -. Vitamin E, Chemotherapy, Oral Mucositis, Voriconazole, Levofloxacin Children and Cancer.
   * Date of search: 01\3\2018
   * Following databases were searched:

     *PubMed database. *Hand searching (Google scholars).

     * The Cochrane Library.

     • The search was limited to English articles only. Electronic and manual searches were performed
     * Inclusion criteria for Articles:

       a. Articles written in English language only. b. Articles including oral mucositis. c. Randomized clinical trials, systematic reviews and meta-analysis.
     * Exclusion criteria for Articles:

       1. Articles including other Vitamin than Vitamin E.
       2. Articles with treatment approaches.

   Methods

   Study setting:
   * The study will be conducted in Department of Pediatric Oncology, National Cancer Institute.
   * Data for this particular study will be collected at Pediatric Department, National Cancer Institute.

   Participants:

   Eligibility criteria:

   Inclusion criteria:

   All children fulfilling the following criteria will be included:

<!-- -->

1. Patients with healthy and intact oral mucosa.
2. Patients diagnosed with Acute Myeloid leukemias for the first time or during consolidation cycle.
3. Both male and female patients undergoing chemotherapy at in and Out patient units of Pediatric Oncology department.
4. Age of patient ranging (6- 18) years old.
5. Legal representatives of patient must be able to read, understand and provide informed consent to participate in the trial.
6. Patients with no history of dental discomfort related to cold or hot food or beverage intake.
7. Patients receiving chemotherapeutic regimen known to cause oral mucositis (e.g. Cytarabine and Etoposide).

Exclusion criteria:

Exclusion criteria included the presence of any of the following:

1. Administration of antiviral or antifungal therapy and/or any other treatment for oral mucositis before enrollment in the study.
2. Presence of advanced or severe periodontitis (pocket depth more than 6mm).
3. Patients who are scheduled for radiotherapy as part of their treatment. Intervention

Diagnosis:

1. Diagnostic chart (Appendix C) will be filled with personal, medical and dental history.
2. The Intraoral examination will be made using mask, gloves, sterile gauze and wooden tongue depressors.
3. Patients who agreed to participate in the study will watch a video explaining how to perform oral hygiene.

   Intervention Group (Vitamin E) - The parents will be instructed to empty the oil contained within 100 IU soft gelatinous capsule which is equivalent to 100 mg of vitamin "E" (Pharco Pharmaceuticals, Egypt).

   - The capsule will be emptied into the child's oral cavity twice daily by piercing it with sterile wrapped needles.

   - Parents will be instructed to wear plastic gloves during these procedures.
   * For older children, the patients will be instructed to chew the vitamin "E" capsule and keep the oil in their mouth for few minutes then swallow it.
   * These procedures will be done on the day of chemotherapy infusion and 5 days after.
   * Follow up for the patient will be done at 7th, 14th and 21st day of chemotherapy infusion.

   Control Group:

   Standard protocol will be used (Voriconazole and Levofloxacin). Criteria for discontinuing intervention In case of any signs of allergy to vitamin E, the treatment will be terminated and the patient will be treated and excluded from the study.

   Strategies to improve adherence to intervention Face to face settings with the patients and their parents to stress on the importance of follow up. This will take place during the study period and during recruitment.

   Participants Timeline:

   Time point Enrollment Allocation Close out 0 7th 14th 21st Diagnostic chart and Intra oral examination X Application of Interventions X Follow up X x X

   Postoperative instructions

<!-- -->

1. Patients are instructed to maintain oral hygiene care as tolerated using soft toothbrush and dental floss.
2. Lip lubrication (Vaseline or Cocoa butter) is instructed to be used.
3. Sugar free gums are advised to enhance oral moistness.
4. Avoidance of certain foods as acidic juices and spicy foods.

   Sample size:

   The aim of this study is to evaluate Prevention of Oral Mucositis After Using Oral Topical Vitamin E Versus Voriconazole and Levofloxacin in Pediatric Cancer Patients Receiving Chemotherapy. According previous researches and books as Isaac and Michael (1995) 10-30 participants will be satisfactory.

   Recruitment strategy:

   Pediatric Cancer patients attending in and Out Pediatric Oncology Units at the National Cancer Institute in Cairo, seeking chemotherapy. Patients will be enrolled in the study if they are compatible with the eligibility criteria.

   Randomization & allocation concealment:

   A) Sequence generation:

   - Computer sequence generated random numbers will be used.

   - Randomization is done by computer software www.random.com.

   - The sequence generates 2 codes (A & B).

   - Each code stands for either intervention or control.

   - The table with the numbers will be with the assistant supervisor.

   B) Allocation concealment mechanism:

   - A telephone call to the assistant supervisor will be done to know the group of the patient.

   C) Implementation:
   * Sequence will be generated by the assistant supervisor and provided through a telephone call.

   Bias:

<!-- -->

1. Selection bias: is reduced by randomization using random number generator and allocation concealment.
2. Performance bias: One operator will perform the trial with a standardized method for all patients.
3. Detection: All outcomes will be detected.
4. Reporting: All outcomes will be reported.

Blinding:

- Blinding for outcome assessor and the statistician

Data management:

Data will be stored on the investigator's personal computer, secured with a password with backup for the data on Google Drive, on hard copy and backup external hard drive.

Monitoring:

The study work results will be monitored regularly by the supervisors.

Statistical method:

Data will be analyzed using IBM SPSS advanced statistics (Statistical Package for Social Sciences), version 24 (SPSS Inc., Chicago, IL). Numerical data will be described as mean and stander deviation or median and range. Categorical data will be described as number and percentage. Data will be explored for normality using Kolmogrov-Smirnv test and Shapiro-Wilk test. Comparisons between two groups for normally distributed numeric variable will be done using the student's test while for non normally distributed numeric variables will be done by the Mann-Whitney U test, Comparisons between categorical variables will be performed using the chi square test A p-value less than or equal to 0.05 will be considered statistically significant. All tests will be two tailed.

Harms:

Vitamin E is considered to have a very low allergic effect and is generally well-tolerated.

Auditing:

Auditing of the study design will be done by the Evidence Based Committee - Faculty of Dentistry - Cairo University.

Research Ethics Approval:

This study protocol and the informed consent form will be reviewed by the Ethics Committee of Scientific Research -National Cancer Institute and Faculty of Dentistry- Cairo University.

Protocol Amendments:

Any modifications to the protocol which may impact the conduct of the study, potential benefit of the patient or may affect patient safety, including changes of study objectives, study design, sample sizes, study procedures, or significant administrative aspect will require a formal amendment to the protocol. Such amendment will be agreed upon by the Council of Pediatric Dentistry and Dental Public Health Department.

Consent and assent:

Researcher will discuss the trial with legal guardian of each participating patient.

* Verbal assent will be taken orally from participating child.
* Written consent will be taken from the legal guardian of each participating child willing to participate in the trial. All consent forms will be translated into Arabic.

Confidentiality:

All study-related information will be stored securely. All participant information will be stored in locked file cabinets in areas with limited access.

Declaration of interests:

The study will be self-funded by investigator and carried out on patients from in or outpatient clinic in Pediatric Cancer Department, National Cancer Institute, Cairo.

Access to data:

Supervisors will be given access to the data sets. All data sets will be password protected.

post-trial care: - Preventive measures as oral hygiene measures will be offered for all participants.

Dissemination policy:

- Study results will be published as partial fulfillment of the requirements for Master degree in Pediatric Dentistry.

* Topics suggested for publication will be circulated to the authors.
* Thesis defense after completion of the study will be done in public with external judges.

ELIGIBILITY:
Inclusion Criteria:

* All children fulfilling the following criteria will be included:

  1. Patients with healthy and intact oral mucosa.
  2. Patients diagnosed with Acute Myeloid leukemias for the first time or during consolidation cycle.
  3. Both male and female patients undergoing chemotherapy at in and Out patient units of Pediatric Oncology department.
  4. Age of patient ranging (6- 18) years old.
  5. Legal representatives of patient must be able to read, understand and provide informed consent to participate in the trial.
  6. Patients with no history of dental discomfort related to cold or hot food or beverage intake.
  7. Patients receiving chemotherapeutic regimen known to cause oral mucositis (e.g. Cytarabine and Etoposide).

Exclusion Criteria:

* Exclusion criteria included the presence of any of the following:

  1. Administration of antiviral or antifungal therapy and/or any other treatment for oral mucositis before enrollment in the study.
  2. Presence of advanced or severe periodontitis (pocket depth more than 6mm).
  3. Patients who are scheduled for radiotherapy as part of their treatment.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Clinical assessment of Oral Mucositis | 5 days
  Oral mucositis WHO Toxicity Scale (Paula Elaine et al., 2016)will be ranked according to WHO classification criteria (Appendix B):
  * Grade 0: No change.
  * Grade 1: Soreness/erythema. • Grade 2: Erythema, and Ulcers; patient can eat solids. • Grade 3: Ulcers; the patient requires liquid diet only. • Grade 4: Oral nourishment is not possible.

CONTACTS AND LOCATIONS:
Locations (1):
- Samah Omer Mekki, Cairo, Egypt